CLINICAL TRIAL: NCT02923271
Title: Promoting Intrafamily Accountability for Reducing Cellphone Use While Driving in Adults and Their Teen Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15-011835
Record Dates: First submitted 2016-10-03; First posted 2016-10-04 (Estimated); Results first posted 2019-08-09 (Actual); Last update posted 2019-08-20 (Actual); Status verified 2019-08

CONDITIONS: Teen Drivers; Motor Vehicle Accidents
Keywords: Driving; Teens; Texting; Cellphone; DriveID; Motor vehicle accident

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Teen-Parent Monitoring Group (Experimental): Cellcontrol DriveID device will automatically turn on when the teen or parent begins driving and will be pre-set to block all calls and text messages when the car is in motion but participants will have the ability to override the blocking. The teen-parent monitoring group involves will send email notifications to the teen when their parent unlocks their phone while driving and vice versa.
  Participants (parents and teens) will self-report information on their individual driving behaviors for the three weeks prior to study enrollment, including how often they report texting while driving and self-report cellphone use. At the end of the study participants will be asked to report feedback about the use the cellphone blocking technology and their perceptions for whether their safety improved using the technology.
  Interventions: Device: CellControl
- Teen Only Monitoring Group (Experimental): Cellcontrol DriveID device will automatically turn on when the teen or parent begins driving and will be pre-set to block all calls and text messages when the car is in motion but participants will have the ability to override the blocking. The teen only group involves parental monitoring of the teen's cellphone use while driving only. The parent will receive an email notification when their teen unlocks their phone while driving. Both parents and teens will drive under the same restrictions, but only the parent is notified of teen cellphone use.
  Participants (parents and teens) will self-report information on their individual driving behaviors for the three weeks prior to study enrollment, including how often they report texting while driving and self-report cellphone use. At the end of the study participants will be asked to report feedback about the use the cellphone blocking technology and their perceptions for whether their safety improved using the technology.
  Interventions: Device: CellControl

INTERVENTIONS:
Device: CellControl — Technology that blocks incoming and outgoing calls and texts. CellControl Drive ID will monitor all cellphone use while driving (without blocking) for 3 weeks during baseline measurement period. During the intervention period (5 weeks) cellphone use will be monitored and blocking of incoming calls and texts will be active.
  Other Names: DriveID

SUMMARY:
Research participants and their parents will be recruited to take part in a randomized control trial. Participants' and their parents' cellphone use will be observed during an initial baseline period. Participants and their parents will then be randomly assigned to one of two conditions: opt-out blocking with parental notification, opt-out blocking with bidirectional notification.

DETAILED DESCRIPTION:
In 2012, 3,328 people were killed and an additional 421,000 were injured in crashes involving a distracted driver. Adults aged greater than 40 years old accounted for 44% of these fatalities. Teen driving behavior is heavily influenced by parental driving behaviors with a recent study showing the proportion of teens that text while driving is 14% higher if they have observed their parents doing the same. The proportion of adults who text while driving has recently surpassed teen rates with a 2013 national poll finding 49% of adult car commuters admit to texting while driving, most stating that they did it out of habit. Based on previous findings, it is unlikely that teens will reduce their texting while driving unless their parents do the same.

The objective of this study is to compare measures of acceptance and feasibility across teen-parent dyads randomized to bidirectional teen-parent (teen monitors parent and parent monitors teen) vs. teen only (parent monitors teen) cellphone use while driving.

Research participants will be recruited to take part in a randomized control trial. Participants' cellphone use will be observed during an initial baseline period. Participants will be randomly assigned to one of two conditions (bidirectional teen-parent monitoring or parental monitoring of the teen only). An exit survey and interview will be administered to both the parent and teen separately at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Both parent and teen will be enrolled together as a pair
* Teen:

  * Is a high school student (age 16 or 17 at start of the study)
  * Holds a valid driver's license
  * Lives in parent/guardian's home
  * Primarily drives one car
  * Drives an average of 4 or more trips per week
  * Has their own iPhone 4S or newer or Android 4.3 or newer smartphone with data plan
  * Admits to texting while driving at least once in the last month
* Parent:

  * Is the parent of a teen driver
  * Drives an average of 4 or more trips per week
  * Primarily drives one car
  * Has their own iPhone 4S or newer or Android 4.3 or newer smartphone with data plan
  * Admits to texting while driving at least once in the last month

Exclusion Criteria:

* Parent and/or teen already uses a smartphone app or hardware device to limit cellphone use while driving

Ages: 16 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 34 (Actual)
Dates: Start 2016-12-07 (Actual); Primary Completion 2017-09-13 (Actual); Study Completion 2017-11-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Catherine McDonald, PhD, RN, Principal Investigator — Children's Hospital of Philadelphia
Locations (2):
- United States (2):
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Teen-Parent Monitoring Group: Cellcontrol DriveID device will automatically turn on when the teen or parent begins driving and will be pre-set to block all calls and text messages when the car is in motion but participants will have the ability to override the blocking. The teen-parent monitoring group involves will send email notifications to the teen when their parent unlocks their phone while driving and vice versa.
  Participants (parents and teens) will self-report information on their individual driving behaviors for the three weeks prior to study enrollment, including how often they report texting while driving and self-report cellphone use. At the end of the study participants will be asked to report feedback about the use the cellphone blocking technology and their perceptions for whether their safety improved using the technology.
  CellControl: Technology that blocks incoming and outgoing calls and texts. CellControl Drive ID will monitor all cellphone use while driving (without blocking) for 3 weeks
- Teen Only Monitoring Group: Cellcontrol DriveID device will automatically turn on when the teen or parent begins driving and will be pre-set to block all calls and text messages when the car is in motion but participants will have the ability to override the blocking. The teen only group involves parental monitoring of the teen's cellphone use while driving only. The parent will receive an email notification when their teen unlocks their phone while driving. Both parents and teens will drive under the same restrictions, but only the parent is notified of teen cellphone use.
  Participants (parents and teens) will self-report information on their individual driving behaviors for the three weeks prior to study enrollment, including how often they report texting while driving and self-report cellphone use. At the end of the study participants will be asked to report feedback about the use the cellphone blocking technology and their perceptions for whether their safety improved using the technology.
  CellControl:
Period: Overall Study
Arm/Group | Teen-Parent Monitoring Group | Teen Only Monitoring Group
Started | 18 | 16
Completed | 10 | 14
Not Completed | 8 | 2

BASELINE CHARACTERISTICS:
Groups:
- Teen Only Monitoring Group: Cellcontrol DriveID device will automatically turn on when teen or parent begins driving blocking. The teen only group involves parental monitoring of the teen's cellphone use while driving only. The parent will receive an email notification when their teen unlocks their phone while driving. Both parents and teens will drive under the same restrictions, but only the parent is notified of teen cellphone use.Participants (parents and teens) will self-report information on their individual driving behaviors for the three weeks prior to study enrollment, including how often they report texting while driving and self-report cellphone use. At the end of the study participants will be asked to report feedback about the use the cellphone blocking technology and their perceptions for whether their safety improved using the technology. CellControl: see other arm
- Total: Total of all reporting groups
Arm/Group | Teen-Parent Monitoring Group | Teen Only Monitoring Group | Total
Number analyzed (Participants) | 18 | 16 | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 9 | 8 | 17
  Between 18 and 65 years | 9 | 8 | 17
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 10 | 25
  Male | 3 | 6 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 0 | 3
  Not Hispanic or Latino | 15 | 16 | 31
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 16 | 14 | 30
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 18 | 16 | 34

OUTCOME MEASURES:

1. Primary Outcome: Change in Number of Cellphone Unlocks Per Hour of Drive Time
Description: Change in number of cellphone unlocks per hour of drive time between baseline and the end of the intervention period
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: Cell phone unlocks per hour
Arm/Group | Teen-Parent Monitoring Group | Teen Only Monitoring Group
Number analyzed (Participants) | 10 | 14
Cell phone unlocks per hour | 0.81 (1.25) | 3.61 (9.32)

2. Secondary Outcome: Change in the Number of Minutes of Phone Use Per Hour of Driving
Description: Change in the number of minutes of phone use per hour of driving between baseline and the end of the intervention
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: Change in the number of minutes of phone
Arm/Group | Teen-Parent Monitoring Group | Teen Only Monitoring Group
Number analyzed (Participants) | 10 | 14
Change in the number of minutes of phone | -4.23 (5.75) | -6.32 (6.71)

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | Teen-Parent Monitoring Group | Teen Only Monitoring Group
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/16
Other Adverse Events (participants affected / at risk) | 0/18 | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-10-06): https://cdn.clinicaltrials.gov/large-docs/71/NCT02923271/Prot_SAP_000.pdf